CLINICAL TRIAL: NCT04241549
Title: A Phase 1 Study of Cusatuzumab Plus Azacitidine in Japanese Patients With Newly Diagnosed Acute Myeloid Leukemia or High-risk Myelodysplastic Syndrome Who Are Not Candidates for Intensive Treatment
Brief Title: A Study of Cusatuzumab Plus Azacitidine in Japanese Participants With Newly Diagnosed Acute Myeloid Leukemia or High-risk Myelodysplastic Syndrome Who Are Not Candidates for Intensive Treatment
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: OncoVerity, Inc. (Industry)
Collaborators: argenx (Industry); Janssen Pharmaceutical K.K. (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: CR108732; 74494550AML1002 (Other: Janssen Pharmaceutical K.K., Japan)
Record Dates: First submitted 2020-01-23; First posted 2020-01-27 (Actual); Last update posted 2023-08-09 (Actual); Status verified 2023-08

CONDITIONS: Leukemia, Myeloid, Acute
MeSH Terms: conditions — Leukemia, Myeloid, Acute | interventions — Azacitidine

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (2):
- Part 1 (Dose Finding): Cusatuzumab + Azacitidine (Experimental): Participants with acute myeloid leukemia (AML) will receive cusatuzumab intravenously (IV) in combination with azacitidine subcutaneously (SC) or IV. The dose levels will be escalated based on the decisions of the Study Evaluation Team (SET) until the recommended Phase 2 Dose (RP2D) has been identified.
  Interventions: Drug: Cusatuzumab; Drug: Azacitidine
- Part 2 (Dose Expansion): Cusatuzumab + Azacitidine (Experimental): Participants with acute myeloid leukemia (AML) and high-risk myelodysplastic syndromes (MDS) will receive cusatuzumab intravenously (IV) at the recommended Phase 2 dose (RP2D) determined in Part 1 in combination with azacitidine subcutaneously (SC) or IV.
  Interventions: Drug: Cusatuzumab; Drug: Azacitidine

INTERVENTIONS:
Drug: Cusatuzumab — Cusatuzumab at a dose 20 milligram per kilogram (mg/kg) once every 2 weeks will be administered intravenously.
  Other Names: JNJ-74494550; ARGX-110
Drug: Azacitidine — Azacitidine at a dose 75 milligram per square meters (mg/m^2) will be administered subcutaneously or intravenously.
  Other Names: VIDAZA

SUMMARY:
The purpose of this study is to determine the recommended Phase 2 dose and evaluate safety profile of cusatuzumab in combination with azacitidine in Japanese participants with treatment naïve acute myeloid leukemia (AML) who are not candidates for intensive treatment.

ELIGIBILITY:
Inclusion Criteria:

* For acute myeloid leukemia (AML) participants: AML according to World Health Organization (WHO) 2016 criteria and fulfilling all of the following criteria:(a) more than or equal to (>=) 75 years of age, or younger participants who are not eligible for or not willing to receive an intensive treatment (including stem cell transplantation) with curative intent and (b) previously untreated AML (except: emergency leukapheresis, low dose of cytarabine and/or hydroxyurea during the screening phase to control hyperleukocytosis but must be discontinued at least one day prior to start of cusatuzumab [Part 1] or azacitidine [Part 2]). All trans retinoic acid (ATRA) treatment for presumed acute promyelocytic leukemia (APL) is permitted but must be discontinued at least 1 day prior to the start of cusatuzumab (Part 1) or azacitidine (Part 2)
* For Myelodysplastic Syndrome (MDS) participants (only for Part 2): MDS according to WHO 2016 criteria and fulfilling all of the following criteria: (a) Not eligible for or not willing to receive allogenic stem cell transplantation,(b) very high or high-risk MDS according to Revised International Prognostic Scoring System (IPSS-R) and (c) previously untreated MDS (except: transfusion and/or cytokine therapy including erythropoietin)
* Eastern Cooperative Oncology Group (ECOG) performance status score of 0, 1 or 2
* Must sign an informed consent form (ICF) indicating that he or she understands the purpose of, and procedures required for, the study and is willing to participate in the study
* A woman of childbearing potential must have a negative highly sensitive serum (beta human chorionic gonadotropin [beta hCG]) or urine pregnancy at screening

Exclusion Criteria:

* Acute promyelocytic leukemia (APL) with t (15;17), or its molecular equivalent promyelocytic leukemia retinoic acid receptor (PML RAR alpha)
* Leukemic involvement or clinical symptoms of leukemic involvement of the central nervous system
* Known allergies, hypersensitivity, or intolerance to cusatuzumab or azacitidine or its excipients (example, mannitol, an excipient of azacitidine)
* Prior treatment with a hypomethylating agent for treatment of AML or MDS
* A diagnosis of other malignancy that requires concurrent nonsurgical treatment

Min Age: 20 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 6 (Actual)
Dates: Start 2020-03-25 (Actual); Primary Completion 2021-07-19 (Actual); Study Completion 2021-07-19 (Actual)

PRIMARY OUTCOMES:
Part 1 and Part 2: Number of Participants with Adverse Events (AEs) and Serious Adverse Events (SAEs) | Up to 3 years
  Number of participants with AEs and SAEs will be reported.
Part 1 and Part 2: Number of Participants with Dose-Limiting Toxicity (DLTs) | Up to 42 days
  Number of participants with DLTs will be reported.
Part 1 and Part 2: Severity of DLT as Assessed by National Cancer Institute Common Terminology Criteria for Adverse Events (NCI-CTCAE) | Up to 42 days
  Severity of DLT as assessed by NCI-CTCAE in participants will be reported.

SECONDARY OUTCOMES:
Part 1 and Part 2: Percentage of Participants with Complete Response (CR) | Up to 9 months
  Percentage of participants with complete response based on response criteria per investigator assessment in participants with acute myeloid leukemia (AML) and myelodysplastic syndrome (MDS) will be reported.
Part 1: Objective Response Rate (ORR) | Up to 6 months
  ORR is defined as percentage of participants with CR, CRh and CRi based on response criteria per investigator assessment in participants with AML.
Part 2: Objective Response Rate (ORR) | Up to 9 months
  ORR is defined as the percentage of participants with CR, partial response (PR) and marrow CR based on response criteria per investigator assessment in participants with MDS.
Part 2: Percentage of Participants with Hematologic Improvement (HI) | Up to 9 months
  Percentage of participants with hematologic improvement will be reported according to response criteria per investigator assessment in participants with MDS.
Part 1 and Part 2: Time to Response | Up to 3 years
  Time to response is defined as time from first dose to achieving the first response of CR, CRh, or CRi in participants with AML and CR, PR or marrow CR in participants with MDS..
Part 1 and Part 2: Duration of Response | Up to 3 years
  Duration of response is defined as time from achieving the first response of CR, CRh, or CRi in participants with AML and CR, PR or marrow CR in participants with MDS to hematologic relapse or death of any cause.
Part 1 and Part 2: Red Blood Cell (RBC) or Platelets Transfusion Independence | Up to 3 years
  Transfusion independence (RBC or platelets) is defined as a period of at least 56 consecutive days with no transfusion between first dose of study drug and the last dose of study drug +30 days.
Part 1 and Part 2: Overall Survival (OS) | Up to 3 years
  OS is defined as the time from initial study intervention administration to death from any cause.
Part 1 and Part 2: Maximum Serum Concentration (Cmax) of Cusatuzumab | Up to 3 years
  Cmax is the maximum observed serum concentration.
Part 1 and Part 2: Serum Trough Concentration (Ctrough) of Cusatuzumab | Up to 3 years
  Ctrough is the serum concentration immediately prior to the next drug administration.

CONTACTS AND LOCATIONS:
Overall Officials: Janssen Pharmaceutical K.K., Japan Clinical Trial, Study Director — Janssen Pharmaceutical K.K.
Locations (5):
- Japan (5):
  - Fukushima Medical University Hospital, Fukushima
  - Gunmaken Saiseikai Maebashi Hospital, Maebashi
  - Osaka City General Hospital, Osaka
  - NTT Medical Center Tokyo, Tokyo
  - University of Fukui Hospital, Yoshida

IPD SHARING:
Plan to Share IPD: Undecided